CLINICAL TRIAL: NCT02398448
Title: In Vitro-In Vivo Relationship Study to Assess the Impact of the In Vitro Dissolution Profile on the Pharmacokinetic Parameters Used to Establish Bioequivalence
Brief Title: IVIVR Assessing PK Parameters Used to Establish Bioequivalence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-101(QCL116986)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zyloprim® 300 mg and three dissolution test formulations (Experimental): Regimen A: Zyloprim® 300 mg; Regimen B: Allopurinol 300 mg; undergranulated, high hardness condition; Regimen C: Allopurinol 300 mg; alternative condition 2; Regimen D: Allopurinol 300 mg; alternative condition 3
  Interventions: Drug: Zyloprim® 300 mg; Drug: Allopurinol 300 mg; undergranulated, high hardness condition; Drug: Allopurinol 300 mg; alternative condition 2; Drug: Allopurinol 300 mg; alternative condition 3

INTERVENTIONS:
Drug: Zyloprim® 300 mg
Drug: Allopurinol 300 mg; undergranulated, high hardness condition — There will be a period for interim analysis after administration of Regimen B to determine the formulation within the process design space that provides the desired in vitro dissolution variant for dosing in the subsequent study period
Drug: Allopurinol 300 mg; alternative condition 2 — There will be a period for interim analysis after administration of Regimen C to determine the formulation within the process design space that provides the desired in vitro dissolution variant for dosing in the subsequent study period
Drug: Allopurinol 300 mg; alternative condition 3

SUMMARY:
The purpose of this study is to determine whether defined and limited changes in in vitro dissolution impact the in vivo pharmacokinetics (PK) and relative bioavailability of allopurinol and the active metabolite oxypurinol.

DETAILED DESCRIPTION:
In this study, a single oral dose of Zyloprim® (300 mg tablet) and 3 separate single oral doses of 300 mg allopurinol test formulations (Regimens B, C and D) will be administered sequentially to each subject on separate occasions. Following the administration of Regimens B and C, there will be a period of interim analysis during which the PK data will be reviewed to determine the formulation within the process design space that provides the desired in vitro dissolution variant for dosing in the subsequent study period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18.0 to 35.0 kg/m2 inclusive, or if outside the range, considered not clinically significant by the Investigator. Must not exceed 40.0 kg/m2.
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Subjects who test positive for the HLA-B*5801 allele.
* Subjects who have received the last dose of an IMP (or treatment with a medical device) within the previous 3 months prior to Day 1 or is currently participating in another study of an IMP (or medical device).
* History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
* Current smokers and those who have smoked within the last 12 months prior to Screening. A breath carbon monoxide reading of greater than 10 ppm at Screening.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator at Screening.
* Clinically significant screening laboratory parameters (biochemistry [AST or ALT > 1.5 × ULN], hematology or urinalysis) as judged by the Investigator (laboratory parameters are listed in Appendix 1).
* Positive drugs of abuse test result during Screening or at Admission (drugs of abuse tests are listed in Appendix 1).
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
* Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the Investigator.
* Evidence of renal impairment at Screening, as indicated by an estimated creatinine clearance of <90 mL/min using the Cockcroft-Gault equation.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator. Hayfever is allowed unless it is active.
* Donation or loss of greater than 400 mL of blood within the previous 3 months prior to Screening.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than up to 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration (See Section 11.4).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
PK profile of Zyloprim® and three dissolution test formulations of allopurinol from plasma | Predose (within 30 minutes before dosing), 15, 30, and 45 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, and 96 hours postdose.
  PK endpoints in terms of maximum observed concentration (Cmax), time of occurrence of maximum observed concentration (Tmax), area under the concentration-time curve (AUClast), area under the concentration-time curve (AUC∞) and apparent terminal half-life (t1/2)

SECONDARY OUTCOMES:
Incidence of Adverse Events | 11 weeks
  Changes in Laboratory, Electrocardiogram and Vital Signs Parameters

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Ruddington, United Kingdom